CLINICAL TRIAL: NCT03591224
Title: A Randomized Controlled Trial of Pharmacogenomic Guided Versus Standard Pharmacist Care to Optimize Antidepressant Drug Therapy in a Community Pharmacy Setting
Brief Title: Pharmacogenomic Testing to Optimize Antidepressant Drug Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John Papastergiou Pharmacy Ltd (Industry)
Collaborators: Green Shield Canada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00025062
Record Dates: First submitted 2018-06-25; First posted 2018-07-19 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Depression; Anxiety; Major Depressive Disorder; Generalized Anxiety Disorder; Mood Disorders
Keywords: pharmacogenetics; pharmacogenomics; antidepressants; pharmacy; pharmacist; community
MeSH Terms: conditions — Depression; Anxiety Disorders; Depressive Disorder, Major; Generalized Anxiety Disorder; Mood Disorders | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Intervention Model Description: Enrolled subjects will be randomly assigned to either the control arm (pharmacist standard of care) or intervention arm (pharmacogenetic guided decision making by the pharmacist) in optimizing antidepressant drug therapy. Randomization is done by the primary investigator who isn't directly involved with patient consultations.
Who Masked: Participant, Care Provider
Masking Description: Patients are not told of their group assignment until the end of the study, at which point they would receive a copy of their pharmacogenetic report. The consulting pharmacist also does not have knowledge of the patient's group assignment in the first encounter for baseline data collection. Group assignment is only revealed to the pharmacist after two weeks when the pharmacogenetic report is available on the Pillcheck online portal. Patients assigned to the control group will have their report appear blank to the pharmacist, whereas the intervention patient group will have their full pharmacogenetic report accessible by the consulting pharmacist. Prescribers are also informed via fax briefly of the study protocol and asked to maintain blinding of their patient's group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Pharmacist optimizing antidepressant therapy using the patient's personalized pharmacogenomic report to make recommendations.
  Interventions: Other: Pharmacogenomic Testing
- Control (Placebo Comparator): Pharmacist optimizing antidepressant therapy based on standard of care
  Interventions: Other: Pharmacist Standard of Care

INTERVENTIONS:
Other: Pharmacogenomic Testing — pharmacogenomic drug response test provides personalized insights on a patient's predicted response to medications based on metabolism
  Other Names: Pillcheck; Geneyouin
  Arms: Intervention
Other: Pharmacist Standard of Care — Pharmacist providing standard of care as per usual practice
  Arms: Control

SUMMARY:
A randomized controlled trial comparing pharmacogenomic guided versus standard pharmacist care to optimize antidepressant drug therapy. This study evaluates the effectiveness of pharmacists utilizing pharmacogenomic testing in the community pharmacy setting to help patients find the most appropriate drug therapy option(s) and minimize the risk of side effects in collaboration with prescribing physicians.

DETAILED DESCRIPTION:
Physicians and pharmacists have long been aware of subtle differences between patients in their responses to medications, but until recently did not have the tools to predict a patient's response to a drug before prescribing it. Many commonly prescribed medications are either ineffective or cause significant side effects for some patients. Individual variation in response to prescription drugs due to genetic factors (pharmacogenetics) is a substantial part of this serious clinical issue. Such variation in patient response ranges from failure to benefit from a drug, to adverse drug reactions, and drug-drug interactions when several drugs are taken at the same time. After years of uncertainty over the value of personalized medicine, recent studies show promising approaches for incorporating pharmacogenetics (PGx) data into routine patient care in order to reduce medication issues due to genetic factors.

Over the last decades, clinical PGx research has made significant progress in defining which genetic variations are important for influencing inter-patient variability in drug response. Evidence-based consensus therapeutic guidelines for multiple drug-gene pairs are available and promoted by the Clinical Pharmacogenetic Implementation Consortium (CPIC). Although the primary focus of PGx testing has been on improving drug selection and dosing, a secondary benefit of testing is the improvement of medication adherence.

GeneYouIn has developed the Pillcheck® drug response test that provides personalized insights on a patient's predicted response to medications. To implement the Pillcheck test, GeneYouIn is working with pharmacists who are adept in understanding pharmacogenetic terminology and can consult with prescribing physicians and patients within current scope of practice. GeneYouIn will provide educational seminars on the latest advances in pharmacogenetics and using the Pillcheck report.

This demonstration project will provide critical education to clinical pharmacists to enable utilization of patients' pharmacogenetic data for evidence-base treatment optimization. The Pillcheck report has been carefully designed to make it easy to interpret and integrate in the clinical pharmacy setting. The study will provide insights on the impact of pharmacogenetics testing on solving Drug Therapy Problems.

The Pillcheck test assesses variations in 14 genes responsible for drug transport and metabolism for over 140 commonly prescribed medications. The Pillcheck report can enable pharmacists to effectively identify Drug Therapy Problems and advise physicians on personalized treatment options thus allowing for more rational medication choices and/or dosing.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed one or more antidepressants
* Diagnosed with major depressive disorder and/or generalized anxiety disorder
* Newly initiated on antidepressant therapy or a recent change in therapy and dissatisfied with therapy.
* Experiencing adverse drug reaction(s) or suboptimal response or dissatisfaction with therapy
* Demonstrated dissatisfaction based on a 9-item prescreening questionnaire. Scoring range from 0='not at all' to 4='very much'. If any scores for Q1-3 on side effects >2, or if any scores for Q4-6 on effectiveness <2, or if any scores for Q7-9 on overall opinion of therapy <2.

[Q1. Side effects interfere with my physical activity, Q2. Side effects interfere with my leisure activities, Q3. Side effects interfere with my daily activities, Q4. The medicine I am taking reduces my symptoms, Q5. I am satisfied with the time it takes for the medicine to start to have an effect, Q6. I feel better now than I did before starting the treatment, Q7.I intend to continue using this treatment, Q8. I feel happy with my treatment, Q9. In general, I feel satisfied with the treatment.]

Exclusion Criteria:

* Patients with poor command of English or who are unable to provide fully informed consent
* Liver transplant patient (cheek swab won't detect liver DNA)
* Non-adherent to prescribed drug therapy due to reasons outside of "not feeling better" (non-medical influencing factors)
* Diagnosis of schizophrenia, bipolar disorder, dementia
* Patients under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment Satisfaction with Medicines Questionnaire (SATMED-Q) - general measure of satisfaction to drug therapy | Change of score from baseline to 6 months
  This scale evaluates patient satisfaction of drug treatment for with any chronic disease. It's a brief, self-administer multidimensional generic questionnaire comprising 17 items. There are six categories of questions assessing satisfaction of (1) drug efficacy, (2) side-effects, (3) convenience of use, (4) medical care, (5) impact on activities of daily living and (6) general satisfaction. Scores of individual items range from 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much. A higher total score is an indication of greater satisfaction with drug therapy. Only scores from the side effects category would be summed as negative values. There is no recommended cutoff score, however is used to monitor the overall satisfaction to treatment over the period of the study.
Patient Health Questionnaire (PHQ-9) - measure/monitor the severity of depression | Change of score from baseline to 6 months
  PHQ-9 is a clinical evidence-based scale used to assess the severity of depression. There are nine diagnostic criteria for major depression based on the Diagnostic and Statistical 4th Ed. (DSM-IV) which are scored '0' (not at all), '1' (several days),'2' more than half the days, '3' (nearly every day). The nine items cover experience of pleasure, feeling down, sleep disruption, energy levels, appetite, feeling a failure, trouble concentrating, speaking slowly or being fidgety and having negative thoughts around suicide or self-harm over the previous 2 weeks. The total sum indicates depression severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe.
Generalized Anxiety Disorder-7 (GAD-7) - measure/monitor the severity of anxiety | Change of score from baseline to 6 months
  Evidence-based questionnaire used to monitor the severity of generalized anxiety. The GAD-7 score is calculated by assigning scores of '0' (not at all), '1' (several days),'2' more than half the days, '3' (nearly every day). Questions assess the tendency of feeling nervous, not being able to stop or control worrying, worrying too much about different things, trouble relaxing, being so restless that it's hard to sit still, becoming easily annoyed or irritable, feeling afraid as if something awful might happen. Total sums of 5, 10, and 15 represent mild, moderate, and severe anxiety, respectively.
Sheehan Disability Scale - measure of functional impairment in work/school, social life, and family life | Change of score from baseline to 6 months
  This scale assesses functional impairment using three 0 to 10 point visual analog scales. This can also be interpreted as percentages. Each of the three scales would have the patient represent how have their symptoms disrupted (1) work/school life, (2) social life, and (3) family life/responsibilities. The points from the 3 scales are summed as a global functional impairment score ranging from 0 (unimpaired) to 30 (highly impaired). There is no recommended cutoff score, however is used to monitor the response to treatment over the period of the study. In general, a score of 5 or greater on any of the three scales is associated with significant functional impairment.

SECONDARY OUTCOMES:
Number of pharmacist identified drug therapy problems | Analysis done at the completion of study (~1 year)
  Total number of Drug Therapy Problems related to antidepressant use identified by the pharmacist include the following types (1) Dose too high/overuse/abuse, (2) Dose too low, (3) Unnecessary drug therapy/duplication, (4) Adverse drug reaction / drug interaction, (5) Requires additional drug therapy, (6) Non-adherence, (7) Inappropriate drug for indication
Prescriber acceptance rate of pharmacist's recommendations | Analysis done at the completion of study (~1 year)
  Percentage of prescriber accepted pharmacist recommendations in the intervention group vs. control group

CONTACTS AND LOCATIONS:
Overall Officials: John Papastergiou, B.Sc.Phm, Principal Investigator — University of Toronto; Wilson Li, B.Sc.Phm, Study Director — John Papastergiou Pharmacy Ltd
Locations (2):
- Canada (2):
  - John Papastergiou Pharmacy Ltd - Store#500, Toronto, Ontario
  - John Papastergiou Pharmacy Ltd - Store#994, Toronto, Ontario

REFERENCES:
- [Background] Rejas J, Ruiz MA, Pardo A, Soto J. Minimally important difference of the Treatment Satisfaction with Medicines Questionnaire (SATMED-Q). BMC Med Res Methodol. 2011 Oct 20;11:142. doi: 10.1186/1471-2288-11-142. PMID 22014277
- [Derived] Papastergiou J, Quilty LC, Li W, Thiruchselvam T, Jain E, Gove P, Mandlsohn L, van den Bemt B, Pojskic N. Pharmacogenomics guided versus standard antidepressant treatment in a community pharmacy setting: A randomized controlled trial. Clin Transl Sci. 2021 Jul;14(4):1359-1368. doi: 10.1111/cts.12986. Epub 2021 Feb 28. PMID 33641259
- See also: Company providing pharmacogenetic testing to optimize drug therapy — https://www.pillcheck.ca/
- See also: Sheehan Disability Scale — http://www.cqaimh.org/pdf/tool_lof_sds.pdf
- See also: PHQ-9 Questionnaire — http://www.cqaimh.org/pdf/tool_phq9.pdf